CLINICAL TRIAL: NCT02660567
Title: The Impacts of Using Amr's Maneuver (Cervical Traction) on Atonic Postpartum Hemorrhage; Multi-centre Randomized Controlled Study
Brief Title: Amr's Maneuver and Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ClinAmygate (Other)
Collaborators: Cairo University (Other); Ain Shams University (Other); October 6 University (Other); National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15127
Record Dates: First submitted 2016-01-19; First posted 2016-01-21 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage; PPH; atonic; new maneuver
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amr Maneuver (Experimental): Active management of third stage plus Amr's maneuver
  Interventions: Procedure: Amr maneuver
- Active management alone (No Intervention): Active management of third stage alone

INTERVENTIONS:
Procedure: Amr maneuver — sustained traction of the anterior and posterior lips of the cervix by ovum forceps downwards and anteriorly until maximum yield for about 90 seconds
  Arms: Amr Maneuver

SUMMARY:
The impacts of using Amr's manoeuvre (cervical traction) on atonic postpartum hemorrhage is a randomized controlled, multi-centre study that aims to compare the incidence of post partum hemorrhage (PPH> 500 ml blood loss) within the first 24 hours of labor after using Amr's maneuver with active management of the third stage versus active management alone

DETAILED DESCRIPTION:
Primary:

Compare the incidence of post partum hemorrhage (PPH> 500 ml blood loss) within the first 24 hours of labor after using Amr's maneuver with active management of the third stage versus active management alone

Secondary:

Comparing:

* The amount of blood loss in each arm of the study
* Hematocrit before and after labor
* Duration from delivery of placenta till discharge from the delivery room

ELIGIBILITY:
Inclusion Criteria:

* All pregnant females aged 18 years or more, candidate for normal vaginal delivery during the period of the study will be included

Exclusion Criteria:

* Women presenting with pre-existing maternal hemorrhagic conditions such as factor 8 or 9 deficiency or Von Willebrand's disease or those who had assisted vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
the incidence of postpartum hemorrhage | 24 hour
  the incidence of post partum hemorrhage (PPH> 500 ml blood loss) within the first 24 hours of labor after using Amr's maneuver with active management of the third stage

CONTACTS AND LOCATIONS:
Overall Officials: Osama Azmy, MD, Principal Investigator — Egypt National Research Centre Reproductive Health Research Department; Emad RH Issak, DM, Study Director — ClinAmygate
Locations (1):
- Cairo University Hospitals (Kasr Al-Aini), Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374
- [Derived] Hamdy A, Azmy O, Lotfy R, Attia AA, Elsherbini MM, Al Sawaf A, Soliman MM, Sharaf MF, Kamel A, Abd El-Raouf MN, Salem S, Rasheed MA, Torky H, Issak ER. Multicenter randomized controlled trial assessing the impact of a cervical traction maneuver (Amr's maneuver) on the incidence of postpartum hemorrhage. Int J Gynaecol Obstet. 2019 Jan;144(1):56-61. doi: 10.1002/ijgo.12687. Epub 2018 Oct 22. PMID 30281778